CLINICAL TRIAL: NCT02768961
Title: Program of Screening, Prevention and Elimination of Hepatitis C in Penitentiary Institutions in Cantabria. JAILFREE-C
Brief Title: Program of Screening, Prevention and Elimination of Hepatitis C in Penitentiary Institutions in Cantabria (JAILFREE-C)
Acronym: JAILFREE-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCG-SOFLDP-2015-01
Record Dates: First submitted 2016-05-02; First posted 2016-05-11 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C
Keywords: sofosbuvir; ledipasvir; ribavirin; prisoner; hepatitis c; prevalence; hepatitis b
MeSH Terms: conditions — Hepatitis C; Hepatitis B | interventions — Sofosbuvir; ledipasvir, sofosbuvir drug combination; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active treatment (Experimental): All HCV chronic infected patients will be treated with oral anti-HCV regimens containing sofosbuvir, ledipasvir (associated or not to ribavirin) according to clinical practice as indicated into the current guidelines (1)
  (1)European Association for Study of Liver (EASL). EASL Recommendations on Treatment of Hepatitis C 2015. J Hepatol. 2015 Jul;63(1):199-236. doi: 10.1016/j.jhep.2015.03.025. Epub 2015 Apr 21. PubMed PMID: 25911336.
  Interventions: Drug: sofosbuvir; Drug: ledipasvir

INTERVENTIONS:
Drug: sofosbuvir — Subjects will be treated according to the current guidelines on HCV treatment taking into account the stage of fibrosis, genotype, previous treatments, etc.
  Sofosbuvir will be used in association with ledipasvir. In some cases, ribavirin can be added to this combination according to current guidelines
  Other Names: Harvoni
Drug: ledipasvir — Subjects will be treated according to the current guidelines on HCV treatment taking into account the stage of fibrosis, genotype, previous treatments, etc.
  Ledipasvir will be used in association with sofosbuvir. In some cases, ribavirin can be added to this combination according to current guidelines
  Other Names: Harvoni

SUMMARY:
The objectives of this study are:

1. To perform a systematic screening and evaluation of the prevalence of infection by hepatitis C virus (HCV), hepatitis B virus (HBV) and human immunodeficiency virus (HIV) in the prison population.
2. To perform an adequate characterization of patients and the characteristics of HCV infection in this population.
3. To evaluate the effectiveness and security in the prison population of an interferon-free antiviral regimen.
4. To evaluate the impact of a strategy of systematic HCV treatment on the rates of persistent infection, reinfection and super-infection in a prison population, in the short, medium and long term.

DETAILED DESCRIPTION:
Background:

Infections caused by hepatitis B, C and HIV viruses represent a serious health problem. The inmate population represents a reservoir with high prevalence of these kind of infections. The completion of a secondary prevention through early detection of infections in early stages, and tertiary prevention by treatment of diagnosed cases, constitutes one of the pillars of the approach to these diseases. This strategy is even more valuable in the inmate population because it can help eliminate a source of spread of these diseases in addition to relieving the burden of disease in this population. In this regard, one of the mandates of the recently adopted National Strategy Plan for the Hepatitis C in Spain emphasizes these strategies.

Finally, a program of this nature is intended as a pilot experience that could be extended to other prison communities at national and European level.

Endpoints

1. - To estimate the prevalence of HBV, HCV and HIV in the inmate population of El Dueso.
2. - To perform a systematic treatment of the inmate population against HCV infection. The treatment will be directed to both, the prevalent population and the new prisoners who enter the prison. The other detected infections will be also treated accordingly.
3. - To carry out a descriptive evaluation of the efficacy and safety of an interferon-free regimen against the HCV infection in this population. This regimen will be mainly based on Sofosbuvir and ledipasvir (± RBV) according to the current clinical practice adopted in the National Strategy Plan for the Hepatitis C.
4. - To evaluate the rates of persistent infection, reinfection and super-infection as defined.

Projected Study Design

The present study is divided in two parts. A transversal and observational one of epidemiological basis aimed to determine the prevalence of viral infections by hepatitis B and C viruses and also by HIV in the inmate population.

In a second prospective phase of follow-up, a systematic treatment of the infected cohort will be carried out in accordance with the current clinical practice adopted in the National Strategy Plan for the Hepatitis C. Data on efficacy, safety and quality of life will be collected throughout the study. Finally, an evaluation of the rates of persistent infection, reinfection and super-infection will be also recorded. Treatment of new admissions throughout the study periods is also contemplated.

Patients and Methods:

Patients:

1. - Epidemiological transversal phase: 435 subjects (the whole inmate population) will be included.
2. - Prospective observational phase: 120 infected patients (taking into account a reported chronic HCV infection prevalence of 20% in the inmate population -data from the latest National Strategic Plan for addressing hepatitis C in the National Health Service "NHS" 2015-) and that it is intended to treat newly infected inmate who enter in prison during the two years of study.

Endpoints:

Primary endpoint: Sustained Virological Response (SVR) at 12 weeks after the end of treatment.

Secondary outcomes: SVR at 4 weeks, Safety issues, Quality of life, Serum prevalence of chronic HCV, HBV infection; re-infection/superinfection rates; cost-effectiveness

Variables:

Variables: HCV status by ELISA; Viral load (PCR) HCV IU / ml (primary), treatment type and duration, serological status of HBV infection; liver stiffness through Fibroscan. QoL variables, ultrasonographic variables. phylogenetic analysis of HCV genome in cases of non-response. costs

Projected Number of Sites (if additional sites, please specify)

1 (El Dueso Penitentiary Centre)

Participating Countries

1 (Spain)

Anticipated First Patient In

2-1-2016

Projected Duration of Enrollment

1 month for the prevalent inmate population. The entry of subjets (new inmates) will be open throughout the study

Projected Duration of Treatment

6 month (8-24 weeks according to patient and virological characteristics).

Study Duration

31 months (1 month enrollment + 6 months of treatment + 24 months observation and final evaluation of reinfections)

ELIGIBILITY:
Inclusion Criteria:

* Epidemiology study: All inmates at the El Dueso Penitentiary Centre including new admissions within the study period.
* Interventional study: All HCV infected patients with detectable viral load (HCV RNA)
* Informed consent signature

Exclusion Criteria:

* Not informed consent signature.
* Pregnant or breastfeeding women
* Hypersensitivity or any temporary or permanent absolute contraindication to either drug that should be prescribed according to clinical and virological characteristics of the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of chronic hepatitis C | 12 months after the beginning of the study.
  Percentage of viremic hepatitis C patients with respect to the whole inmate population
Percentage of Participants with Sustained Virological Response | 12 weeks after the end of treatment
  Percentage of Participants with Sustained Virological Response (undetectable viral load) at this point

SECONDARY OUTCOMES:
Adverse events | 4 weeks after the start of treatment
  Presence and type of adverse events at this point.
Adverse events | 8 weeks after the start of treatment
  Presence and type of adverse events at this point.
Adverse events | 12 weeks after the start of treatment
  Presence and type of adverse events at this point.
Adverse events | 24 weeks after the start of treatment
  Presence and type of adverse events at this point.
Percentage of Participants with Sustained Virological Response | 4 weeks after the end of treatment
  Percentage of Participants with Sustained Virological Response (undetectable viral load) at this point
HCV seroprevalence | baseline
  Presence of anti-HCV at baseline
HBV seroprevalence | baseline
  Presence of HBsAg seropositivity
HIV seroprevalence | baseline
  Presence of anti-HIV at baseline
Chronic HCV infection prevalence | baseline
  Detectable HCV RNA viral load at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Javier Crespo García, MDPhD, Study Director — Head of Gastroenterology and Hepatology at Hospital Universitario Marqués de Valdecilla; Carmen Cobo Pelayo, MD, Principal Investigator — Ministerio del Interior. Secretaría General de Instituciones Penitenciarias
Locations (1):
- Penitentiary "El Dueso". Cantabria. Spain, Santoña, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Association for Study of Liver. EASL Recommendations on Treatment of Hepatitis C 2015. J Hepatol. 2015 Jul;63(1):199-236. doi: 10.1016/j.jhep.2015.03.025. Epub 2015 Apr 21. No abstract available. PMID 25911336
- [Background] Rice JP, Burnett D, Tsotsis H, Lindstrom MJ, Cornett DD, Voermans P, Sawyer J, Striker R, Lucey MR. Comparison of hepatitis C virus treatment between incarcerated and community patients. Hepatology. 2012 Oct;56(4):1252-60. doi: 10.1002/hep.25770. PMID 22505121